CLINICAL TRIAL: NCT03443973
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Efficacy, and Safety Study of Gantenerumab in Patients With Early (Prodromal to Mild) Alzheimer's Disease
Brief Title: Safety and Efficacy Study of Gantenerumab in Participants With Early Alzheimer's Disease (AD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision to terminate development of Gantenerumab for treatment of prodromal/mild/early stage Alzheimer's disease following results of a pre-planned analysis of the safety and efficacy of Gant in Graduate I&II (WN29922/WN39658).
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WN39658; 2017-001365-24 (EudraCT Number)
Record Dates: First submitted 2018-02-19; First posted 2018-02-23 (Actual); Results first posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — gantenerumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gantenerumab (Experimental): Gantenerumab will be administered as SC injections with gradual uptitration.
  Interventions: Drug: Gantenerumab
- Placebo (Placebo Comparator): Placebo will be administered as SC injections with gradual uptitration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gantenerumab — Gantenerumab will be administered as per the schedule specified in the respective arm.
  Other Names: RO4909832
  Arms: Gantenerumab
Drug: Placebo — Placebo matching to gantenerumab will be administered as per the schedule specified in the respective arm.
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled, parallel group study will evaluate the efficacy and safety of gantenerumab versus placebo in participants with early (prodromal to mild) AD. All participants must show evidence of beta-amyloid pathology. Eligible participants will be randomized 1:1 to receive either subcutaneous (SC) injection of gantenerumab or placebo. The primary efficacy assessment will be performed at the end of the double blind period at week 116. Participants will then be offered to enter into an open-label extension (OLE). Participants not willing to go to the OLE will participate in a long term follow-up period for up to 50 weeks after the last gantenerumab dose.

ELIGIBILITY:
Key Inclusion criteria:

* Meets National Institute on Aging/Alzheimer's Association (NIAAA) core clinical criteria for probable AD dementia or prodromal AD (consistent with the NIAAA diagnostic criteria and guidelines for mild cognitive impairment)
* Evidence of the AD pathological process, as confirmed by CSF tau/A-beta42or amyloid PET scan
* Demonstrated abnormal memory function
* MMSE score greater than or equal to 22 (≥ 22)
* Clinical dementia rating-global score (CDR-GS) of 0.5 or 1.0
* Availability of a reliable study partner who accepts to participate in study procedures throughout the 2 years duration of study
* If receiving symptomatic AD medications, the dosing regimen must have been stable for 3 months prior to screening and until randomization
* For enrollment in the China extension, patients must have residence in mainland China, Hong Kong, or Taiwan and be of Chinese ancestry
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods

Key Exclusion criteria:

* Any evidence of a condition other than AD that may affect cognition
* History of schizophrenia, schizoaffective disorder, major depression, or bipolar disorder
* History or presence of clinically evident systemic vascular disease that in the opinion of the investigator has the potential to affect cognitive function
* History or presence of clinically evident cerebrovascular disease
* History or presence of posterior reversible encephalopathy syndrome
* History or presence of any stroke with clinical symptoms within the past 12 months, or documented history within the last 6 months of an acute event that is consistent with a transient ischemic attack
* History of severe, clinically significant CNS trauma
* History or presence of intracranial mass (e.g., glioma, meningioma) that could potentially impair cognition
* Presence of infections that affect brain function or history of infections that resulted in neurologic sequelae
* History or presence of systemic autoimmune disorders that potentially cause progressive neurologic disease with associated cognitive deficits
* At risk for suicide in the opinion of the investigator
* Alcohol and/or substance abuse or dependants in past 2 years
* Relevant brain hemorrhage, bleeding disorder and cerebrovascular abnormalities
* Any contraindications to brain MRI
* Unstable or clinically significant cardiovascular, kidney or liver disease
* Uncontrolled hypertension
* Unstable or clinically significant cardiovascular disease
* Abnormal thyroid function
* Patients with evidence of folic acid deficiency

Exclusion for Open-Label Extension (OLE):

* Discontinued from study treatment during the double-blind treatment period
* Received any other investigational medication during the double-blind treatment period or after the end of double-blind treatment
* Participation in the OLE deemed inappropriate by the investigator
* Presence of ARIA-E findings at the Week 116 MRI scan

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 975 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (155):
- United States (47):
  - Banner Alzheimer?s Institute, Phoenix, Arizona
  - Barrow Neurological Institute, Phoenix, Arizona
  - Banner Sun Health Research Insitute, Sun City, Arizona
  - Health Initiatives Research, PLLC, Fayetteville, Arkansas
  - Fullerton Neurology and Headache Center, Fullerton, California
  - Neurology Center of North Orange County, Fullerton, California
  - Irvine Center for Clinical Research, Irvine, California
  - Desert Valley Research, Redlands, California
  - Southern California Research LLC, Simi Valley, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Accel Research Sites - CRU Tampa, Bradenton, Florida
  - ClinCloud, LLC, Maitland, Florida
  - Optimus U Corp, Miami, Florida
  - Allied Biomedical Research Institute, Inc, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - Infinity Clinical Research, LLC, Sunrise, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Rush Alzheimer's Disease Cntr., Chicago, Illinois
  - American Health Network Institute, LLC, Avon, Indiana
  - Brigham and Womens Hospital; Center for Alzheimer Research & Treatment, Boston, Massachusetts
  - ActivMed Practices and Research, Haverhill, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - Missouri Memory Center, Bolivar, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center; Dept of Neurological Sciences, Omaha, Nebraska
  - Cleveland Clinic Lou Ruvo; Center for Brain Research, Las Vegas, Nevada
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - AD-CARE, University of Rochester Medical Center, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Behavioral Health Research, Charlotte, North Carolina
  - Alzheimer's Memory Center, Matthews, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Neuro-Behavioral Clinical Research, Inc., Canton, Ohio
  - Cleveland Clinic; Cleveland Lou Ruvo Center for Brain Health ? Neurological Institute, Cleveland, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Summit Research Network Inc., Portland, Oregon
  - Texas Neurology PA, Dallas, Texas
  - Kerwin Medical Center, Dallas, Texas
  - Alzheimers Disease & Memory Disorders Center; Department of Neurology Baylor College of Medicine, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
- Argentina (7):
  - Hospital Italiano, Buenos Aires
  - Universidad Maimonides, Caba
  - Instituto Geriatrico Nuestra Señora de las Nieves, Capital Federal
  - Instituto Kremer, Córdoba
  - CEN Centro Especializado en Neurociencias, Córdoba
  - Instituto de Neurociencias San Agustín S.A., La Plata
  - Fundacion Scherbovsky, Mendoza
- Belgium (3):
  - AZ Sint Blasius (Dendermonde), Dendermonde
  - UZ Gent, Ghent
  - Jessa Zkh (Campus Virga Jesse), Hasselt
- Chile (3):
  - Psicomed Estudios Médicos, Antofagasta
  - Biomedica Research Group, Santiago
  - Especialidades Medicas LYS, Santiago
- Clinical Hospital Centre Zagreb;Clinic for Neurology, Zagreb, Croatia
- Denmark (3):
  - Aarhus Universitetshospital; Neurologisk Afd. F, Demensklinikken, Aarhus N
  - Rigshospitalet, Hukommelsesklinikken, København Ø
  - Svendborg Sygehus; Neurologisk afdeling N, Demensklinik Fyn, Svendborg
- Finland (2):
  - Terveystalo Ruoholahti, Helsinki
  - University of Eastern Finland, Kuopio
- Japan (16):
  - Yachiyo Hospital, Aichi
  - Nagoya Ekisaikai Hospital, Aichi
  - National Center for Geriatrics and Gerontology, Aichi
  - Fukuoka University Hospital, Fukuoka
  - National Hospital Organization Hiroshima-Nishi Medical Center, Hiroshima
  - Hyogo Prefectural HarimaHimeji General Medical Center, Hyōgo
  - Tsukazaki Hospital, Hyōgo
  - Matsui Dietary and Dementia Clinic, Hyōgo
  - Kagawa Prefectural Central Hospital, Kagawa
  - Rakuwakai Otowa Hospital, Kyoto
  - Uji Takeda Hospital, Kyoto
  - Rijikai Medical Corporation Katayama Medical Clinic, Okayama
  - Kishiwada Tokushukai Hospital, Osaka
  - National Hospital Organization Hizen Psychiatric Medical Center, Saga
  - Medical corporation Ichiekai Itsuki Hospital, Tokushima
  - Tokushima Hospital, Tokushima
- Mexico (4):
  - Mexico Centre for Clinical Research, Mexico City, Mexico CITY (federal District)
  - Hospital Universitario Dr Jose Eleuterio Gonzalez UANL; Depto.de NeurologíaPta.BajaConsulta, Monterrey, Nuevo León
  - AVIX Investigación Clínica S.C, Monterrey, Nuevo León
  - Hospital Angeles Culiacan; Neurociencias, Culiacán, Sinaloa
- Brain Research Center B.V, Amsterdam, Netherlands
- Poland (10):
  - O?rodek Badawczo-Naukowo-Dydaktyczny Chorób Ot?piennych w ?cinawie, ?cinawa
  - Podlaskie Centrum Psychogeriatrii, Bia?ystok
  - NZOZ Vitamed, Bydgoszcz
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - Neurologiczny NZOZ Centrum Leczenia SM; Osrodek Badan Klinicznych, Plewiska
  - NEURO-CARE Sp. z o.o. Sp. Komandytowa, Siemianowice ?l?skie
  - Senior Sp. Z O.O. Poradnia Psychogeriatryczna, Sopot
  - mMED Maciej Czarnecki, Warsaw
  - Pratia S.A., Warsaw
  - NZOZ WCA, Wroc?aw
- Portugal (5):
  - Hospital Prof. Dr. Fernando Fonseca; Servico de Neurologia, Amadora
  - Hospital de Braga; Servico de Neurologia, Braga
  - HUC; Servico de Neurologia, Coimbra
  - Hospital da Senhora da Oliveira-Guimarães; Serviço de Neurologia, Guimarães
  - Hospital Geral de Santo Antonio; Servico de Neurologia, Porto
- Puerto Rico (2):
  - Santa Cruz Behavioral PSC, Bayamón
  - University of Puerto Rico - Medical Science Campus; Internal Medicine, San Juan
- Singapore (2):
  - National University Hospital (NUH); Neuroscience, Singapore
  - National Neuroscience Institute; Neurology, Singapore
- South Korea (12):
  - Dong-A University Hospital, Busan
  - Myongji Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Hanyang University Seoul Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Ewha Womans University Hospital (Seoul), Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
- Spain (15):
  - Hospital General Universitario de Elche; Servicio de Neurología, Elche, Alicante
  - Hospital Mutua De Terrasa; Servicio de Neurologia, Terrassa, Barcelona
  - Hospital Virgen del Puerto. Servicio de Neurología, Plasencia, Caceres
  - Policlínica Guipuzcoa; Servicio de Neurología, Donostia / San Sebastian, Guipuzcoa
  - Hospital Universitario de Santa Maria; Servicio de Neurología, Lleida, Lerida
  - Hospital Quiron de Madrid; Servicio de Neurologia, Pozuelo de Alarcón, Madrid
  - Clinica Universitaria de Navarra; Servicio de Neurología, Pamplona, Navarre
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - CAE OROITU; Servicio de Neurología, Getxo, Vizcaya
  - Hospital del Mar; Servicio de Neurologia, Barcelona
  - Fundación ACE; Servicio de Neurología, Barcelona
  - Universitario de La Princesa; Servicio de Neurología, Madrid
  - Hospital Victoria Eugenia; Servico Neurología, Seville
  - Hospital Universitario la Fe; Servicio de Neurologia, Valencia
  - Complejo Asistencial de Zamora; Servicio Psiquiatria, Zamora
- Sweden (3):
  - Skånes Universitetssjukhus Malmö, Minneskliniken, Malmo
  - Sahlgrenska Academy University,Neuroscience and Physiology;Departmt of Psychiatry and Neurochemistry, Mölndal
  - KAROLINSKA UNI HOSPITAL, HUDDINGE; Mottagning Kognitiv Forskning, M54, Stockholm
- Turkey (Türkiye) (3):
  - Istanbul University Istanbul School of Medicine; Neurology, Istanbul
  - Bezmialem Vakif Univ Medical, Istanbul
  - Ondokuz Mayis Univ. Med. Fac.; Neurology, Samsun
- United Kingdom (16):
  - Royal Cornhill Hospital; OAP Directorate, Aberdeen
  - The Rice Centre; Royal United Hospital, Bath
  - Re-Cognition, Birmingham
  - The Fritchie Centre, Charlton Lane Centre, Charlon Lane, Leckhampton; The Fritchie Centre, Cheltenham
  - Surrey and Borders NHS Foundation Trust; Brain Science Research Unit, Chertsey
  - Sussex Partnership NHS Foundation Trust; Cognitive Treatment and Research unit, Crowborough
  - Ninewells Hospital, Dundee
  - Queen Elizabeth University Hospital; Clinical Research Facility, Glasgow
  - St George's Hospital, London
  - RE:Cognition Health, London
  - Charing Cross Hospital, London
  - Campus for Ageing and Vitality, Newcastle
  - John Radcliffe Hospital, Oxford
  - Royal Preston Hospital, Preston
  - Royal Hallamshire Hospital Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - University Southampton NHS Foundation Trust; Wessex Neurologica Centre, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Chandler JM, Lansdall CJ, Ye W, McDougall F, Belger M, Toth B, Mi X, Sink KM, Atkins AS. The Alzheimer's Disease Cooperative Study - Activities of Daily Living dependence score: revision and validation of an algorithm evaluating patient dependence across the spectrum of AD severity. J Prev Alzheimers Dis. 2025 Sep;12(8):100261. doi: 10.1016/j.tjpad.2025.100261. Epub 2025 Jul 1. PMID 40603145
- [Derived] Asada T, Thanasopoulou A, Delmar P, Wojtowicz J, Smith J, Yoshiyama Y, Yokoi K, Watanabe C, Isozaki M, Ozaki R, Ishida T, Tatsuda H, Tamaoka A. Japanese participant data from three gantenerumab trials in early Alzheimer's disease. Alzheimers Dement. 2025 Apr;21(4):e70192. doi: 10.1002/alz.70192. PMID 40302041
- [Derived] Bittner T, Tonietto M, Klein G, Belusov A, Illiano V, Voyle N, Delmar P, Scelsi MA, Gobbi S, Silvestri E, Barakovic M, Napolitano A, Galli C, Abaei M, Blennow K, Barkhof F. Biomarker treatment effects in two phase 3 trials of gantenerumab. Alzheimers Dement. 2025 Feb;21(2):e14414. doi: 10.1002/alz.14414. Epub 2025 Jan 30. PMID 39887500
- [Derived] Salloway S, Wojtowicz J, Voyle N, Lane CA, Klein G, Lyons M, Rossomanno S, Mazzo F, Bullain S, Barkhof F, Bittner T, Schneider A, Grundman M, Aldea R, Boada M, Smith J, Doody R. Amyloid-Related Imaging Abnormalities (ARIA) in Clinical Trials of Gantenerumab in Early Alzheimer Disease. JAMA Neurol. 2025 Jan 1;82(1):19-29. doi: 10.1001/jamaneurol.2024.3937. PMID 39556389
- [Derived] Bateman RJ, Smith J, Donohue MC, Delmar P, Abbas R, Salloway S, Wojtowicz J, Blennow K, Bittner T, Black SE, Klein G, Boada M, Grimmer T, Tamaoka A, Perry RJ, Turner RS, Watson D, Woodward M, Thanasopoulou A, Lane C, Baudler M, Fox NC, Cummings JL, Fontoura P, Doody RS; GRADUATE I and II Investigators and the Gantenerumab Study Group. Two Phase 3 Trials of Gantenerumab in Early Alzheimer's Disease. N Engl J Med. 2023 Nov 16;389(20):1862-1876. doi: 10.1056/NEJMoa2304430. PMID 37966285

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study across 151 investigative sites in 18 countries from 22 August 2018 to 28 November 2022.
Pre-assignment Details: A total of 975 participants with early (prodromal to mild) Alzheimer's Disease (AD) were randomized to either the gantenerumab (n=498) or placebo arm (n=477) to enter the double-blind treatment (DBT) period.
Groups:
- Placebo: DBT: Participants received, gantenerumab matching placebo, subcutaneous (SC) injections, every four weeks (Q4W) up to Week 36 and then every two weeks (Q2W) up to Week 114 of the DBT period.
- Gantenerumab: DBT: Participants received gantenerumab, SC injections with gradual up-titration starting at a dose of 120 milligrams (mg), Q4W for 3 doses, followed by 255 mg, Q4W for 3 doses, and 510 mg, Q4W for 3 doses. Following this, from Week 36 onwards, participants received gantenerumab, SC injections, at a dose of 510 mg, Q2W up to Week 114 of the DBT period.
- Placebo (DBT) to Gantenerumab: Open-label Extension (OLE): Participants who received gantenerumab matching placebo in the DBT period received gantenerumab SC injections with gradual up titration starting at a dose of 120 mg, Q4W for 3 doses, followed by 255 mg, Q4W for 3 doses, and then at a dose of 510 mg, Q4W up to Week 34 of the OLE period. To maintain the blind to previous treatment assignment, participants received Q2W, SC injections, with alternate doses containing gantenerumab matching placebo.
- Gantenerumab (DBT) to Gantenerumab: OLE: Participants who received gantenerumab in the DBT period continued receiving gantenerumab, SC injections, 510 mg, Q2W up to Week 34 of the OLE period.
Period: Double-blind Treatment Period
Arm/Group | Placebo: DBT | Gantenerumab: DBT | Placebo (DBT) to Gantenerumab: Open-label Extension (OLE) | Gantenerumab (DBT) to Gantenerumab: OLE
Started | 477 | 498 | 0 | 0
Safety-evaluable Set (Safety-evaluable set included all participants randomized during the global phase, who received at least one dose of study drug. In DBT period, three participants randomized to placebo arm received at least one dose of gantenerumab and were considered in the gantenerumab arm for safety evaluable set.) | 474 | 501 | 0 | 0
Completed | 397 | 372 | 0 | 0
Not Completed | 80 | 126 | 0 | 0
Not completed — Adverse Event | 5 | 19 | 0 | 0
Not completed — Death | 5 | 7 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Reason Not Specified | 9 | 11 | 0 | 0
Not completed — Physician Decision | 5 | 6 | 0 | 0
Not completed — Protocol Deviation | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 54 | 79 | 0 | 0
Period: Open-label Extension Period
Arm/Group | Placebo: DBT | Gantenerumab: DBT | Placebo (DBT) to Gantenerumab: Open-label Extension (OLE) | Gantenerumab (DBT) to Gantenerumab: OLE
Started | 0 (Participants who completed the DBT Period were given the option to enroll in the OLE Period to receive gantenerumab.) | 0 (Participants who completed the DBT Period were given the option to enroll in the OLE Period to receive gantenerumab.) | 13 (13 Participants who completed the DBT Period enrolled into the OLE Period.) | 14 (14 Participants who completed the DBT Period enrolled into the OLE Period.)
Completed | 0 | 0 | 8 | 13
Not Completed | 0 | 0 | 5 | 1
Not completed — Reason Not Specified | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all participants randomized during the global phase, who received at least one dose of study drug.
Groups:
- Placebo: DBT: Participants received, gantenerumab matching placebo, SC injections, Q4W up to Week 36 and then Q2W up to Week 114 of the DBT period.
- Gantenerumab: DBT: Participants received gantenerumab, SC injections with gradual up-titration starting at a dose of 120 mg, Q4W for 3 doses, followed by 255 mg, Q4W for 3 doses, and 510 mg, Q4W for 3 doses. Following this, from Week 36 onwards, participants received gantenerumab, SC injections, at a dose of 510 mg, Q2W up to Week 114 of the DBT period.
- Total: Total of all reporting groups
Arm/Group | Placebo: DBT | Gantenerumab: DBT | Total
Number analyzed (Participants) | 477 | 498 | 975
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (7.4) | 71.6 (7.8) | 71.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 285 | 288 | 573
  Male | 192 | 210 | 402
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 119 | 112 | 231
  Not Hispanic or Latino | 358 | 386 | 744
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13 | 13 | 26
  Asian | 75 | 56 | 131
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 385 | 424 | 809
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Clinical Dementia Rating-Sum of Boxes (CDR-SB) [Mean (Standard Deviation); unit: score on a scale] — CDR was derived through semi-structured interview with participant and appropriate informant. It rated impairment across 6 domains: memory,orientation,judgment,and problem solving,community affairs,home and hobbies, and personal care on a 5-point scale for which 0=no impairment, 0.5=questionable impairment, and 1, 2, and 3=mild, moderate, severe impairment respectively. The CDR-SB is based on summing each of the domain box scores with total score ranging from 0-18 with higher scores reflecting greater cognitive and functional impairment. Population: ITT analysis set included all participants randomized during the global phase, who received at least one dose of study drug. Overall number analyzed is the number of participants with data available for analysis.
  score on a scale
    number analyzed (Participants) | 477 | 497 | 974
    (all) | 3.52 (1.54) | 3.67 (1.61) | 3.60 (1.58)

OUTCOME MEASURES:

1. Primary Outcome: DBT Period: Change From Baseline to Week 116 in Global Outcome, as Measured by CDR-SB
Description: CDR was derived through semi-structured interview with the participant and an appropriate informant, and it rated impairment across six domains: memory, orientation, judgment, and problem solving, community affairs, home and hobbies, and personal care on a 5-point scale for which 0=no impairment, 0.5=questionable impairment, and 1, 2, and 3=mild, moderate, and severe impairment, respectively. The CDR-SB is based on summing each of the domain box scores with total score ranging from 0-18 with higher scores reflecting greater cognitive and functional impairment. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 116
Population: ITT analysis set included all participants randomized during the global phase, who received at least one dose of study drug. Overall number analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo: DBT | Gantenerumab: DBT
Number analyzed (Participants) | 477 | 497
score on a scale | 3.01 (0.15) | 2.82 (0.14)
Statistical Analysis 1: Comparison: Placebo: DBT vs Gantenerumab: DBT; Change from Baseline was calculated based on ANCOVA analysis model which included the following covariates and stratification factors =Treatment + Baseline (BL) + Geographic Region + Disease Stage + AD Medication at BL + Apolipoprotein E, Allele e4 (APOE e4) + Baseline ADAS COG13 + Baseline Alzheimer Disease Cooperative Study Group-Activities of Daily Living (ADCS-ADL); Test type: Superiority; p = 0.2998, ANCOVA; Difference in Adjusted mean = -0.19, 95% CI 2-sided [-0.55 to 0.17], Standard Error of Mean 0.18

2. Primary Outcome: OLE Period: Number of Participants With Adverse Events (AEs)
Description: An adverse event is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution.
Time Frame: From day of first dose in OLE period up to 14 weeks after the last OLE dose (up to 48 weeks)
Population: OLE safety-evaluable set included all participants randomized during the global enrollment phase who received at least one dose of study drug and who entered the OLE period.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (DBT) to Gantenerumab: Open-label Extension (OLE) | Gantenerumab (DBT) to Gantenerumab: OLE
Number analyzed (Participants) | 13 | 14
Participants | 8 | 6

3. Primary Outcome: OLE Period: Number of Participants With Post-baseline Suicidal Ideation or Suicidal Behavior as Measured Using Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS=assessment tool used to assess lifetime suicidality of a participant (at baseline) as well as any new instances of suicidality (C-SSRS since last visit). Structured interview prompts recollection of suicidal ideation, including intensity of ideation, behavior, & attempts with actual/potential lethality. Categories have binary responses (yes/no) & include Wish to be Dead; Non-specific Active Suicidal Thoughts; Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Active Suicidal Ideation with Specific Plan and Intent, Preparatory Acts and Behavior; Aborted Attempt; Interrupted Attempt; Actual Attempt (non-fatal); Completed Suicide. Suicidal ideation/behavior is indicated by a "yes" answer to any of the listed categories. Score of 0 is assigned if no suicide risk is present. Score of 1 or higher= suicidal ideation or behavior. Categories with non-zero values are only reported here.
Time Frame: From day of first dose in OLE period up to 14 weeks after the last OLE dose (up to 48 weeks)
Population: OLE safety-evaluable set included all participants randomized during the global enrollment phase who received at least one dose of study drug and who entered the OLE period. Overall number analyzed is the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (DBT) to Gantenerumab: Open-label Extension (OLE) | Gantenerumab (DBT) to Gantenerumab: OLE
Number analyzed (Participants) | 12 | 13
Participants
  Suicidal Ideation: Passive | 1 | 0
  Suicidal Ideation: Active-Method, but no Intent or Plan | 1 | 0
  Suicidal Ideation: No Event | 10 | 13
  Suicidal Behavior: No event | 12 | 13
  Self-injurious Behavior Without Suicidal Intent: No event | 12 | 13

4. Primary Outcome: OLE Period : Number of Participants With Amyloid-Related Imaging Abnormalities-Haemosiderin Deposition (ARIA-H) Confirmed by MRI
Description: ARIA are an identified risk with anti-amyloid antibodies, including gantenerumab. These changes can be identified on brain MRI. ARIA-H (H for hemosiderosis) are small foci of signal loss observed on MRI sequences sensitive for paramagnetic tissue properties and comprise cerebral microbleeds (small foci of bleeding in the brain parenchyma) and leptomeningeal hemosiderosis (small foci of bleeding on the surface of the brain). These changes also occur sporadically in AD.
Time Frame: From day of first dose in OLE period up to 14 weeks after the last OLE dose (up to 48 weeks)
Population: MRI Safety-evaluable analysis set included all participants in the Safety-evaluable analysis set who had at least one post-baseline safety MRI scan.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (DBT) to Gantenerumab: Open-label Extension (OLE) | Gantenerumab (DBT) to Gantenerumab: OLE
Number analyzed (Participants) | 13 | 14
Participants | 2 | 1

5. Primary Outcome: OLE Period: Number of Participants With Amyloid-Related Imaging Abnormalities-Edema (ARIA-E) Confirmed by Magnetic Resonance Imaging (MRI)
Description: ARIA are an identified risk with anti-amyloid antibodies, including gantenerumab. These changes can be identified on brain MRI. In ARIA-E, (E for oedema or effusion), oedema can be seen in different areas of the brain on MRI, representing fluid leakage into the brain parenchyma or sulcal spaces.
Time Frame: From day of first dose in OLE period up to 14 weeks after the last OLE dose (up to 48 weeks)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (DBT) to Gantenerumab: Open-label Extension (OLE) | Gantenerumab (DBT) to Gantenerumab: OLE
Number analyzed (Participants) | 13 | 14
Participants | 0 | 1

6. Primary Outcome: OLE Period: Number of Participants With Injection-Site Reactions
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product or other protocol-imposed intervention, regardless of attribution. Local injection reactions (or injection site reactions) are defined as AEs related to the injection site that occur during or within 24 hours after study drug administration that are judged to be related to the study drug injection.
Time Frame: From day of first dose in OLE period up to 14 weeks after the last OLE dose (up to 48 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (DBT) to Gantenerumab: Open-label Extension (OLE) | Gantenerumab (DBT) to Gantenerumab: OLE
Number analyzed (Participants) | 13 | 14
Participants | 0 | 1

7. Secondary Outcome: DBT Period: Change From Baseline to Week 116 in Alzheimer Disease Assessment Scale-Cognition Subscale 13 (ADAS-Cog13) Score
Description: The ADAS-Cog13 total score includes all of the items in the ADAS-Cog11 in addition to delayed word recall and the number cancellation. For the ADAS-cog 13 the range is 0-85 (score range for Delayed Word Recall [DWR] score is 0-10 and for Number Cancellation [NC] is 0-5, thus the score is ADAS-cog 11[0-70] plus the scores for DWR and NC). A higher score indicates worse performance. A negative change from baseline indicates improvement in cognitive function.
Time Frame: Baseline, Week 116
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo: DBT | Gantenerumab: DBT
Number analyzed (Participants) | 475 | 491
score on a scale | 7.94 (0.49) | 6.66 (0.42)
Statistical Analysis 1: Comparison: Placebo: DBT vs Gantenerumab: DBT; Change from BL was calculated based on ANCOVA analysis model which included the following covariates and stratification factors = Treatment + Baseline + Geographical Region + Disease Stage + AD Medication at BL + APOE e4; Test type: Superiority; p = 0.0273, ANCOVA; Difference in adjusted mean = -1.28, 95% CI 2-sided [-2.41 to -0.14], Standard Error of Mean 0.58

8. Secondary Outcome: DBT Period: Change From Baseline to Week 116 in Alzheimer's Disease Cooperative Study- Activities of Daily Living (ADCS-ADL) Total Score
Description: ADCS-ADL is a 23-item rater-administered, observer-reported outcome (ObsRO) that captures a participant's ability to perform basic activities of daily living (e.g., eating and toileting) and more complex ADL or instrumental activities of daily living (iADL, e.g., using the telephone, managing finances, preparing a meal). Total score ranges from 0-78, with higher scores reflecting better functioning. A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 116
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo: DBT | Gantenerumab: DBT
Number analyzed (Participants) | 475 | 496
score on a scale | -9.26 (0.62) | -8.44 (0.58)
Statistical Analysis 1: Comparison: Placebo: DBT vs Gantenerumab: DBT; Change from BL was calculated based on ANCOVA analysis model which included the following covariates and stratification factors = Treatment + Baseline + Region + Disease Stage + AD Medication at BL + APOE e4; Test type: Superiority; p = 0.2918, ANCOVA; Difference in adjusted mean = 0.82, 95% CI 2-sided [-0.70 to 2.34], Standard Error of Mean 0.78

9. Secondary Outcome: DBT Period: Change From Baseline to Week 116 in Functional Activities Questionnaire (FAQ) Score
Description: FAQ is a rater-administered ObsRO (informant-based measure) that measures a participant's functional ability to perform complex higher-order activities. The observer provides performance ratings of the target person on ten complex higher-order activities. Total score that ranges from 0-30, with higher scores reflecting greater functional impairment. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 116
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo: DBT | Gantenerumab: DBT
Number analyzed (Participants) | 476 | 496
score on a scale | 6.72 (0.33) | 5.86 (0.31)
Statistical Analysis 1: Comparison: Placebo: DBT vs Gantenerumab: DBT; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.0438, ANCOVA; Difference in adjusted mean = -0.86, 95% CI 2-sided [-1.70 to -0.02], Standard Error of Mean 0.43

10. Secondary Outcome: DBT Period: Change From Baseline to Week 116 in Mini-Mental State Examination (MMSE) Total Score
Description: MMSE is a rater-administered performance-based outcome (PerfO) that includes a set of standardized questions used to evaluate possible cognitive impairment and help stage the severity level of this impairment. The questions target six areas: orientation, registration, attention, short-term recall, language, and constructional praxis/visuospatial abilities. Total score ranges from 0-30, with lower scores indicating greater impairment. A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 116
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo: DBT | Gantenerumab: DBT
Number analyzed (Participants) | 477 | 497
score on a scale | -4.53 (0.22) | -4.00 (0.20)
Statistical Analysis 1: Comparison: Placebo: DBT vs Gantenerumab: DBT; Change from Baseline was calculated based on ANCOVA analysis model which included the following covariates and stratification factors =Treatment + Baseline + Geographic Region + Disease Stage + AD Medication at BL + APOE e4; Test type: Superiority; p = 0.0566, ANCOVA; Difference in adjusted mean = 0.52, 95% CI 2-sided [-0.01 to 1.06], Standard Error of Mean 0.27

11. Secondary Outcome: DBT Period: Change From Baseline to Week 116 in Alzheimer Disease Assessment Scale-Cognition Subscale 11 (ADAS-Cog11) Score
Description: The ADAS-Cog11 was designed to measure cognitive symptom change in participants with Alzheimer's Disease (AD) and consisted of 11 tasks. The standard 11 items (and corresponding score range) were: word recall (0-10), commands (0-5), constructional praxis (0-5), naming objects and fingers (0-5), ideational praxis (0-5), orientation (0-8), word recognition (0-12), spoken language ability (0-5), comprehension of spoken language (0-5), word-finding difficulty (0-5), and remembering test instructions (0-5). The test included 7 performance items and 4 clinician-rated items. The ADAS-Cog11 total score was the sum of all 11 individual items, with a total score ranging from 0 (no impairment) to 70 (severe impairment). Higher scores indicated more severe cognitive impairment. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 116
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo: DBT | Gantenerumab: DBT
Number analyzed (Participants) | 475 | 491
score on a scale | 6.97 (0.46) | 5.77 (0.38)
Statistical Analysis 1: Comparison: Placebo: DBT vs Gantenerumab: DBT; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.0260, ANCOVA; Difference in adjusted mean = -1.19, 95% CI 2-sided [-2.24 to -0.14], Standard Error of Mean 0.53

12. Secondary Outcome: DBT Period: Change From Baseline to Week 116 in Verbal Fluency Task (VFT) Score
Description: VFT is a rater administered PerfO that measures speed and flexibility of verbal thought with a total score that ranges from 0-99 (lower scores indicating lower performance). A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 116
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo: DBT | Gantenerumab: DBT
Number analyzed (Participants) | 477 | 497
score on a scale | -2.68 (0.22) | -2.71 (0.21)
Statistical Analysis 1: Comparison: Placebo: DBT vs Gantenerumab: DBT; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.9086, ANCOVA; Difference in adjusted mean = -0.03, 95% CI 2-sided [-0.59 to 0.52], Standard Error of Mean 0.28

13. Secondary Outcome: DBT Period: Change From Baseline to Week 116 in the Coding (Digit Symbol Substitution Test [DSST]) Subtest
Description: Coding, also called DSST is a rater administered PerfO that measures speed of processing and associative memory with a total score that ranges from 0-135 (lower scores indicating lower performance). The DSST was adapted from the Wechsler Adult Intelligence Scale. The 120-second version of the test was used in this study. Positive change from baseline indicates improvement.
Time Frame: Baseline, Week 116
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo: DBT | Gantenerumab: DBT
Number analyzed (Participants) | 475 | 497
score on a scale | -6.90 (0.59) | -5.49 (0.55)
Statistical Analysis 1: Comparison: Placebo: DBT vs Gantenerumab: DBT; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.0629, ANCOVA; Difference in adjusted mean = 1.41, 95% CI 2-sided [-0.08 to 2.90], Standard Error of Mean 0.76

14. Secondary Outcome: DBT Period: Change From Baseline to Week 116 in Alzheimer's Disease Cooperative Study-Instrumental Activities of Daily Living (ADCS-iADL) Instrumental Score
Description: The ADCS-iADL measures activities such as using the telephone, shopping and preparing a meal. The ADCS-iADL consists of 16 questions with a score range of 0 to 56 where a higher score represents better function. Positive change from baseline indicates improvement.
Time Frame: Baseline, Week 116
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo: DBT | Gantenerumab: DBT
Number analyzed (Participants) | 475 | 496
score on a scale | -8.22 (0.53) | -7.43 (0.49)
Statistical Analysis 1: Comparison: Placebo: DBT vs Gantenerumab: DBT; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.2348, ANCOVA; Difference in adjusted mean = 0.79, 95% CI 2-sided [-0.51 to 2.09], Standard Error of Mean 0.66

15. Secondary Outcome: DBT Period: Number of Participants With AEs
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution.
Time Frame: From Day 1 up to 14 weeks after the last dose of blinded study drug (up to 128 weeks)
Population: Safety-evaluable set included all participants randomized during the global phase, who received at least one dose of study drug. In the DBT period, three participants randomized to placebo arm received at least one dose of gantenerumab and were considered in the gantenerumab arm for safety evaluable set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: DBT | Gantenerumab: DBT
Number analyzed (Participants) | 474 | 501
Participants | 409 | 451

16. Secondary Outcome: DBT Period: Number of Participants With Post-baseline Suicidal Ideation or Suicidal Behavior as Measured Using C-SSRS
Description: as for outcome 3
Time Frame: From Day 1 up to 14 weeks after the last dose of blinded study drug (up to 128 weeks)
Population: Safety-evaluable set included all participants randomized during the global phase, who received at least one dose of study drug. In the DBT period, three participants randomized to placebo arm received at least one dose of gantenerumab and were considered in the gantenerumab arm for safety evaluable set. Overall number analyzed is the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: DBT | Gantenerumab: DBT
Number analyzed (Participants) | 464 | 483
Participants
  Suicidal Ideation: Passive | 20 | 12
  Suicidal Ideation: Active-Nonspecific | 4 | 2
  Suicidal Ideation: Active-Method, But No Intent or Plan | 2 | 2
  Suicidal Ideation: Active-Method and Intent, But No Plan | 1 | 1
  Suicidal Ideation: Active-Method, Intent, and Plan | 0 | 2
  Suicidal Ideation: No Event | 437 | 464
  Suicidal Behavior: No Event | 464 | 483
  Self-injurious Behavior, No Suicidal Intent | 0 | 2
  Self-injurious Behavior Without Suicidal Intent: No Event | 464 | 481

17. Secondary Outcome: DBT Period: Number of Participants With ARIA-E Confirmed by MRI
Description: as for outcome 5
Time Frame: From Day 1 up to 14 weeks after the last dose of blinded study drug (up to 128 weeks)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: DBT | Gantenerumab: DBT
Number analyzed (Participants) | 470 | 496
Participants | 18 | 128

18. Secondary Outcome: DBT Period: Number of Participants With ARIA-H Confirmed by MRI
Description: as for outcome 4
Time Frame: From Day 1 up to 14 weeks after the last dose of blinded study drug (up to 128 weeks)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: DBT | Gantenerumab: DBT
Number analyzed (Participants) | 470 | 496
Participants | 57 | 109

19. Secondary Outcome: DBT Period: Number of Participants With Injection-Site Reactions
Description: as for outcome 6
Time Frame: From Day 1 up to 14 weeks after the last dose of blinded study drug (up to 128 weeks)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: DBT | Gantenerumab: DBT
Number analyzed (Participants) | 474 | 501
Participants | 31 | 75

20. Secondary Outcome: DBT Period: Number of Participants With Anti-Drug Antibodies (ADA) to Gantenerumab
Description: The number of participants with positive results for ADA against gantenerumab at any of the post-baseline assessment time-points were reported. Participant with an ADA assay result from at least one post-baseline sample was defined as a post-baseline evaluable participant. Treatment Emergent ADA = A participant with a negative or missing baseline ADA result(s) and at least one positive post-baseline ADA result.
Time Frame: From Day 1 up to 14 weeks after the last dose of blinded study drug (up to 128 weeks)
Population: ADA-evaluable analysis set included participants who received at least one dose of study drug and who provided at least one post-baseline ADA sample. In the DBT period, three participants randomized to placebo arm received at least one dose of gantenerumab and were considered in the gantenerumab arm. As pre-specified in the protocol of study WN42171, ADA data for studies WN29922 and WN39658 from the OLE period will be reported in the results of study WN42171 (NCT04374253).
Measure: Count of Participants; unit: Participants
Arm/Group | Gantenerumab: DBT
Number analyzed (Participants) | 501
Participants | 12

21. Secondary Outcome: Change From Baseline to Week 116 in Brain Amyloid Load as Measured by Amyloid Positron Emission Tomography (PET) Scan in a Subset of Participants
Description: Brain amyloid load over time was assessed using [18F] florbetaben or [18F] flutemetamol tracers. These are PET radioligand selective to amyloid. Amyloid PET burden was measured in a composite region of interest (ROI) by using standardized uptake value ratio (SUVR) mapped to the centiloid scale. The weighted composite target region are composed of (both left and right side): frontal lobe, parietal lobe, temporal lobe lateral, cingulum posterior and anterior cingulate gyrus. The reference region used to normalize the composite region was the whole cerebellum. The centiloid scale anchor points are 0 and 100, where 0 represents a high-certainty amyloid negative scan and 100 represents the amount of global amyloid deposition found in a typical AD scan.
Time Frame: Baseline, Week 116
Population: Amyloid-PET-modified-ITT (mITT) included all participants in the ITT analysis set who participated in the Amyloid PET sub-study and who had at least one Amyloid PET scan with a valid quantitative measurement performed with either florbetaben or flutemetamol and who did not withdraw from the Amyloid PET substudy before randomization. Overall number analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo: DBT | Gantenerumab: DBT
Number analyzed (Participants) | 44 | 40
score on a scale | 8.46 (2.768) | -48.00 (2.845)
Statistical Analysis 1: Comparison: Placebo: DBT vs Gantenerumab: DBT; Change from BL was calculated based on mixed-effect model of repeated measure which included the following covariates and stratification factors = Baseline + APOE e4 status + Type of Tracer + Analysis Visit + Treatment + Treatment*Analysis Visit + Analysis Visit*Baseline; Test type: Superiority; p < .0001, Mixed Model for Repeated Measures; Difference in adjusted means = -56.46, 95% CI 2-sided [-64.36 to -48.56], Standard Error of Mean 3.976

22. Secondary Outcome: Change From Baseline to Week 116 in Brain Tau Load, as Measured by Tau PET Scan in a Subset of Participants
Description: Change in tau load= how much neurofibrillary tau pathology is present in brain assessed by PET Scan. Tau PET radioligand used was [18F] GTP1. Tau load was measured using SUVR in 4 composite target ROIs: Temporal target region included (both left & right)=anterior &posterior superior temporal gyrus, posterior temporal lobe, fusiform gyrus, &middle &inferior temporal gyrus; Medial temporal region excluding hippocampus included (both left & right): amygdala, parahippocampus & anterior medial & lateral temporal lobe; Frontal lobe (both left & right) & Parietal lobe (both left & right). Inferior cerebellar grey matter=reference region for calculating SUVRs for 4 target regions. Tau-PET-mITT analysis set=all participants in ITT analysis set who participated in Tau PET sub-study & had at least one Tau PET scan with valid quantitative measurement & who did not withdraw from Tau PET substudy before randomization. Overall number analyzed=number of participants with data available for analysis.
Time Frame: Baseline, Week 116
Population: As pre-specified in protocol/SAP single tau PET substudy analyzed participants from 2 studies i.e. WN29922 (NCT03444870) & WN39658 (NCT03443973), hence data for Tau PET was analyzed at pooled level of WN29922 &WN39658. These studies had identical study design &enrolled an Early AD population. Tau PET analysis was planned in a subset of participants, to get an optimum sample size for analysis, it was pre-planned to conduct one tau PET substudy for participants willing to consent to the procedure.
Measure: Mean (Standard Error); unit: SUVR
Arm/Group | Placebo: DBT | Gantenerumab: DBT
Number analyzed (Participants) | 29 | 48
SUVR
  ROI: Temporal Composite Region | 0.12 (0.018) | 0.13 (0.014)
  ROI: Medial Temporal Composite Region [not including the Hippocampus] | 0.08 (0.014) | 0.09 (0.011)
  ROI: Frontal Lobe | 0.08 (0.012) | 0.08 (0.009)
  ROI: Parietal Lobe | 0.09 (0.020) | 0.09 (0.016)
Statistical Analysis 1: Comparison: Placebo: DBT vs Gantenerumab: DBT; Temporal Composite Region: Change from BL was calculated based on mixed-effect model of repeated measure which included the following covariates and stratification factors = Baseline + APOE e4 status + Study + Analysis Visit + Treatment + Treatment*Analysis Visit + Analysis Visit*Baseline; Test type: Superiority; p = 0.7816, Mixed Model for Repeated Measures; Difference in adjusted mean = 0.01, 95% CI 2-sided [-0.04 to 0.05], Standard Error of Mean 0.023
Statistical Analysis 2: Comparison: Placebo: DBT vs Gantenerumab: DBT; Medial Temporal Composite Region: Change from BL was calculated based on mixed-effect model of repeated measure which included the following covariates and stratification factors = Baseline + APOE e4 status + Study + Analysis Visit + Treatment + Treatment*Analysis Visit + Analysis Visit*Baseline; Test type: Superiority; p = 0.6203, Mixed Model for Repeated Measures; Difference in adjusted means = 0.01, 95% CI 2-sided [-0.03 to 0.05], Standard Error of Mean 0.018
Statistical Analysis 3: Comparison: Placebo: DBT vs Gantenerumab: DBT; Frontal Lobe: Change from BL was calculated based on mixed-effect model of repeated measure which included the following covariates and stratification factors = Baseline + APOE e4 status + Study + Analysis Visit + Treatment + Treatment*Analysis Visit + Analysis Visit*Baseline; Test type: Superiority; p = 0.7754, Mixed Model for Repeated Measures; Difference in adjusted means = 0.00, 95% CI 2-sided [-0.03 to 0.03], Standard Error of Mean 0.015
Statistical Analysis 4: Comparison: Placebo: DBT vs Gantenerumab: DBT; Parietal Lobe: Change from BL was calculated based on mixed-effect model of repeated measure which included the following covariates and stratification factors = Baseline + APOE e4 status + Study + Analysis Visit + Treatment + Treatment*Analysis Visit + Analysis Visit*Baseline; Test type: Superiority; p = 0.9022, Mixed Model for Repeated Measures; Difference in adjusted means = 0.00, 95% CI 2-sided [-0.05 to 0.05], Standard Error of Mean 0.026

23. Secondary Outcome: DBT Period: Percent Change From Baseline to Week 116 in Cerebrospinal Fluid (CSF) Marker of Disease in a Subset of Participants - Neurofilament Light Chain (NFL)
Description: NFL is a neuronal cytoplasmic protein highly expressed in large, myelinated axons. Its levels increase in CSF and blood proportionally to the degree of axonal damage in a variety of neurological disorders, including AD.
Time Frame: Baseline, Week 116
Population: CSF modified ITT analysis set included all participants in the ITT analysis set who had at least one valid quantitative CSF measurement. Overall number analyzed is the number of participants with data available for analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change in NFL
Arm/Group | Placebo: DBT | Gantenerumab: DBT
Number analyzed (Participants) | 72 | 74
percent change in NFL | 25.5 [15.83 to 35.97] | 8.9 [0.60 to 17.83]
Statistical Analysis 1: Comparison: Placebo: DBT vs Gantenerumab: DBT; Test type: Superiority; p = 0.014, ANCOVA; Percent Difference in Geometric Mean = -13.2, 95% CI 2-sided [-22.51 to -2.87]

24. Secondary Outcome: DBT Period: Percent Change From Baseline to Week 116 in CSF Marker of Disease in a Subset of Participants - Neurogranin
Time Frame: Baseline, Week 116
Population: as for outcome 23
Measure: Geometric Mean (95% Confidence Interval); unit: percent change in neurogranin
Arm/Group | Placebo: DBT | Gantenerumab: DBT
Number analyzed (Participants) | 72 | 72
percent change in neurogranin | -6.1 [-11.99 to 0.12] | -19.6 [-24.66 to -14.30]
Statistical Analysis 1: Comparison: Placebo: DBT vs Gantenerumab: DBT; Test type: Superiority; p < 0.001, ANCOVA; Percent Difference in Geometric Mean = -14.4, 95% CI 2-sided [-21.88 to -6.21]

25. Secondary Outcome: DBT Period: Percent Change From Baseline to Week 116 in CSF Marker of Disease in a Subset of Participants - Total Tau (tTau)
Description: CSF biomarker tTau has been considered as a general marker of neurodegeneration. An elevation in levels of tau, as well as specific pTau species, is thought to be a marker for progressive cellular degeneration in AD.
Time Frame: Baseline, Week 116
Population: as for outcome 23
Measure: Geometric Mean (95% Confidence Interval); unit: percent change in tTau
Arm/Group | Placebo: DBT | Gantenerumab: DBT
Number analyzed (Participants) | 72 | 71
percent change in tTau | 1.8 [-4.46 to 8.45] | -16.4 [-21.55 to -10.87]
Statistical Analysis 1: Comparison: Placebo: DBT vs Gantenerumab: DBT; Test type: Superiority; p < 0.001, ANCOVA; Percent Difference in Geometric Mean = -17.8, 95% CI 2-sided [-24.92 to -10.11]

26. Secondary Outcome: DBT Period: Percent Change From Baseline to Week 116 in CSF Marker of Disease in a Subset of Participants - Phosphorylated Tau (pTau-181)
Description: CSF phospho-tau is an indicator of neuronal injury and neurodegeneration. CSF biomarker tTau has been considered as a general marker of neurodegeneration. An elevation in levels of pTau species, is thought to be a marker for progressive cellular degeneration in AD.
Time Frame: Baseline, Week 116
Population: as for outcome 23
Measure: Geometric Mean (95% Confidence Interval); unit: percent change in pTau-181
Arm/Group | Placebo: DBT | Gantenerumab: DBT
Number analyzed (Participants) | 71 | 70
percent change in pTau-181 | 0.1 [-6.50 to 7.16] | -20.9 [-26.17 to -15.31]
Statistical Analysis 1: Comparison: Placebo: DBT vs Gantenerumab: DBT; Test type: Superiority; p < 0.001, ANCOVA; Percent Difference in Geometric Mean = -21.0, 95% CI 2-sided [-28.29 to -12.97]

27. Other Pre Specified Outcome: Plasma Concentration of Gantenerumab
Time Frame: Pre-dose on Days 1, Weeks 24, 52 and 76; Post-dose on Day 4, Weeks 41, 103, and 115
Population: Pharmacokinetic(PK)-evaluable analysis set included participants who received at least one dose of study drug and who provided at least one valid post-baseline PK sample.
Arm/Group | Gantenerumab: DBT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: DBT Period: From Day 1 up to 14 weeks after the last dose of blinded study drug (up to 128 weeks); OLE Period: From day of first dose in OLE period up to 14 weeks after the last OLE dose (up to 48 weeks) All cause mortality: DBT: Day 1 up to the end of study (up to approximately 164 weeks); OLE period: From OLE Day 1 up to the end of the study (up to approx. 86 weeks)
Description: All-cause mortality was reported based on ITT analysis set=all randomized participants.
  SAEs & other AEs reported based on safety-evaluable set=all participants randomized during global phase & received at least one dose of study drug. 3 participants randomized to placebo received at least one dose of gantenerumab and were represented in gantenerumab arm; OLE safety set=all participants randomized during global enrollment phase who received at least one dose of study drug & entered OLE period.
Groups:
- Placebo (DBT) to Gantenerumab: OLE: Participants who received gantenerumab matching placebo in the DBT period received gantenerumab SC injections with gradual up titration starting at a dose of 120 mg, Q4W for 3 doses, followed by 255 mg, Q4W for 3 doses, and then at a dose of 510 mg, Q4W up to Week 34 of the OLE period. To maintain the blind to previous treatment assignment, participants received Q2W, SC injections, with alternate doses containing gantenerumab matching placebo.
Arm/Group | Placebo: DBT | Gantenerumab: DBT | Placebo (DBT) to Gantenerumab: OLE | Gantenerumab (DBT) to Gantenerumab: OLE
All-Cause Mortality (participants affected / at risk) | 5/477 | 7/498 | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 63/474 | 61/501 | 1/13 | 0/14
Other Adverse Events (participants affected / at risk) | 296/474 | 358/501 | 8/13 | 6/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo: DBT (N=474) | Gantenerumab: DBT (N=501) | Placebo (DBT) to Gantenerumab: OLE (N=13) | Gantenerumab (DBT) to Gantenerumab: OLE (N=14)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asymptomatic COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Avulsion fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Focal dyscognitive seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vertebrobasilar stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delusion (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo: DBT (N=474) | Gantenerumab: DBT (N=501) | Placebo (DBT) to Gantenerumab: OLE (N=13) | Gantenerumab (DBT) to Gantenerumab: OLE (N=14)
Arrhythmia (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 15 (16) | 11 (12) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 25 (33) | 39 (44) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 13 (20) | 22 (38) | 1 (1) | 0 (0)
Fatigue (General disorders) | 12 (15) | 15 (17) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 31 (58) | 75 (319) | 0 (0) | 1 (5)
COVID-19 (Infections and infestations) | 30 (31) | 36 (36) | 0 (0) | 1 (1)
Dacryocystitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Groin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 49 (62) | 45 (53) | 1 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 5 (7) | 4 (4) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 5 (5) | 8 (8) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 24 (26) | 29 (38) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 26 (38) | 32 (34) | 0 (0) | 1 (1)
Bone fissure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 47 (58) | 47 (74) | 2 (3) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 7 (7) | 6 (6) | 1 (1) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 9 (12) | 5 (8) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 9 (10) | 10 (15) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Blood pressure diastolic decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 42 (49) | 39 (47) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 32 (39) | 29 (33) | 1 (1) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 (27) | 15 (18) | 0 (0) | 0 (0)
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 2 (2) | 33 (35) | 0 (0) | 0 (0)
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 12 (15) | 114 (162) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 4 (5) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 29 (36) | 39 (54) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 50 (64) | 64 (118) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 9 (9) | 14 (17) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 22 (23) | 26 (31) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 5 (6) | 13 (14) | 1 (1) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (6) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 35 (40) | 34 (38) | 2 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/73/NCT03443973/Prot_002.pdf
  • Statistical Analysis Plan (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/73/NCT03443973/SAP_003.pdf